CLINICAL TRIAL: NCT05936372
Title: Study Protocol to Examine the Effects of Acute Exercise on Motor Learning and Brain Activity in Children With Developmental Coordination Disorder (ExLe-Brain-DCD)
Brief Title: Effects of Acute Exercise on Motor Learning and Brain Activity in Children With DCD
Acronym: ExLeBrainDCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Nacional d'Educacio Fisica de Catalunya (Other)
Collaborators: ICFO - The Institute of Photonic Sciences (Unknown); Ministerio de Ciencia e Innovación, Spain (Other Government); University of Stuttgart (Other); The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Albert Busquets Faciaben, Principal Investigator, Institut Nacional d'Educacio Fisica de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PID2020-120453RB-I00; PID2020-120453RB-I00 (Other Grant/Funding Number: Ministerio de Ciencia e Innovación de España)
Record Dates: First submitted 2023-06-09; First posted 2023-07-07 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Developmental Coordination Disorder
Keywords: Visuomotor adaptation; Attention; Physical exercise; Functional near-infrared spectroscopy (fNIRS); Cortical activation; Prefrontal cortex; Children
MeSH Terms: conditions — Motor Skills Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EX-TD (Experimental): Typical developed children that perform acute exercise prior to the learning task
  Interventions: Behavioral: Acute intense aerobic exercise
- CON-TD (No Intervention): Typical developed children that not perform acute exercise prior to the learning task
- EX-DCD (Experimental): Children with developmental coordination disorder (DCD) that perform acute exercise prior to the learning task
  Interventions: Behavioral: Acute intense aerobic exercise
- CON-DCD (No Intervention): Children with developmental coordination disorder (DCD) that not perform acute exercise prior to the learning task

INTERVENTIONS:
Behavioral: Acute intense aerobic exercise — The acute intense aerobic exercise bout (iE) will consist of a 13-minute 20-meter shuttle run. During this exercise bout two speeds, based on a percentage of the estimated maximal oxygen consumption (VO2max), will be combined: a fast-paced speed (fast: 85% of VO2max) and a slow-paced speed (slow: 60% VO2max). A total of 3 series of 3 min of the fast-paced speed will be carried interspersed with 2 series of 2 min of the slow-paced speed. Prior to the iE start, a warm-up protocol consisting of 2 min slow and 1 min fast will be done with the objective to familiarize participants with the iE speeds. A 5-minute rest period will be guaranteed before starting the iE. Transition time between iE and the rotational visuomotor adaptation task (rVMA) will be 4 min.
  Arms: EX-DCD; EX-TD

SUMMARY:
The aim of this study is to investigate the impact of an acute intense physical exercise bout on the learning ability of children with typical motor development (TD) and children with developmental coordination disorder (DCD). The effects will be studied during the learning and in the short- (1 hour), medium- (24 hours), and long-terms (7 days) after the initial learning. Participants will be divided into 4 groups: children with typical development who will exercise (EX-TD), children with developmental coordination disorder who will exercise (EX-DCD), children with typical development who will not exercise (CON-TD), and children with developmental coordination disorder who will not exercise (CON-DCD). Participants will be enrolled for 4 different sessions:

Session 1: First, participants will do a test to asses their cognitive ability and their height and weight will be measured. Then, participants will run a race test to assess their level of physical condition and to calculate high and moderate intensities of the exercise bout. The test will consist of running from one side to the other of a 20 m long track, while following the rhythm set by a sound.

Session 2: at least 48 hours after the first one, the participants will do an exercise bout running from side to side of a 20 m long track alternating high and moderate intensities during 13 min. The members of the control groups (CON-TD and CON-DCD) will not perform this exercise and, instead, will remain at rest for a time equivalent to the exercise of the other groups. On the other hand, participants will perform a learning task involving hand-eye coordination, in which participants will control the movements of a circle on a computer screen using a joystick. The objective of this task will be to move the circle to target points that will appear on the screen with the maximum accuracy and speed possible. Participants will be asked to practice this task for approximately 8 min. Then, after a 1-hour rest period, the participants will be asked to perform the learning task again (only 3.5 min) to check the level of retention of the initial learning. A headcap will be adjusted on the head of the participants during the motor task performance to measure the activity of the brain through infrared light.

Sessions 3 and 4: participants will complete two retention tests of the learning task (one in each session) 24 hours and 7 days after the second session, respectively. Participants will also wear the headcap for the brain activity measurements.

ELIGIBILITY:
Inclusion Criteria:

* Movement assessment battery for children - second edition (MABC-2) score: developmental coordination disorder (DCD) group score <15% and typically developed (TD) group score >25%
* An average or better cognitive ability tested through the Test of Nonverbal Intelligence version 4 (TONI-4)
* A parent-report history to confirm that, according to the child's pediatrician, motor difficulties showed by their child cannot be explained by any other neurological, developmental, and/or severe psychosocial problem. Comorbid attention deficit hyperactivity disorder, attention deficit disorder, and dyslexia will be acceptable in order to better represent the DCD population since data population-based studies suggest that almost 40% of the children with DCD have combined problems related to learning and/or attentional disorders.

Exclusion Criteria:

* Participant health status do not allow hem/her to participate in physical activities (Physical Activity Readiness Questionnaire, PAR-Q)
* Other comorbidities than attention deficit hyperactivity disorder, attention deficit disorder, and/or dyslexia
* Reported neurological, developmental, and/or severe psychosocial problem that could explain the motor development problem
* Participant that takes medication that could affect results
* Uncorrected 20/20 vision

Ages: 90 Months to 126 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
initial directional error | 0, 1, and 24 hours, and 7 days
  Initial directional error (IDE) will be calculated as the absolute angular difference between the ideal trajectory, a linear vector from the center to the target, and the early real trajectory, defined by the linear vector from the center to the cursor position at the time of 80 ms after movement onset.
root mean square error | 0, 1, and 24 hours, and 7 days
  Root mean square error (RMSE) will be calculated to represent the straightness of the movement between the ideal trajectory and the real joystick trajectory.
initial rate of learning | 0, 1, and 24 hours, and 7 days
  The initial rate of learning (RL) will be computed as the first derivative of the first half of the function and evaluated at epoch 1 for both error variables initial directional error (RL-IDE) and root mean square error (RL-RMSE).
relative oxyhemoglobin concentration ([02Hb]) in the ventrolateral prefrontal cortex | 0, 1, and 24 hours, and 7 days
  Neural activation of each cortical area will be expressed as a relative increase of oxyhemoglobin concentration ([02Hb]) measured by functional near-infrared spectroscopy (fNIRS).
relative oxyhemoglobin concentration ([02Hb]) in the dorsolateral prefrontal cortex | 0, 1, and 24 hours, and 7 days
  Neural activation of each cortical area will be expressed as a relative increase of oxyhemoglobin concentration ([02Hb]) measured by functional near-infrared spectroscopy (fNIRS).
relative deoxyhemoglobin concentration ([HHb]) in the ventrolateral prefrontal cortex | 0, 1, and 24 hours, and 7 days
  Neural activation of each cortical area will be expressed as a relative decrease of deoxyhemoglobin concentration ([HHb]) measured by functional near-infrared spectroscopy (fNIRS).
relative deoxyhemoglobin concentration ([HHb]) in the dorsolateral prefrontal cortex | 0, 1, and 24 hours, and 7 days
  Neural activation of each cortical area will be expressed as a relative decrease of deoxyhemoglobin concentration ([HHb]) measured by functional near-infrared spectroscopy (fNIRS).

SECONDARY OUTCOMES:
movement time | 0, 1, and 24 hours, and 7 days
  Time spend moving the cursor from its initial position to its final position
travel distance | 0, 1, and 24 hours, and 7 days
  Displacement of the cursor from its initial position to its final position
reaction time | 0, 1, and 24 hours, and 7 days
  Reaction time will be defined as the time between target appearance and movement onset.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Busquets Faciaben, PhD, Principal Investigator — Institut Nacional d'Educació Física de Catalunya; Rosa M Angulo Barroso, PhD, Principal Investigator — Institut Nacional d'Educació Física de Catalunya
Locations (3):
- Spain (3):
  - Escola Bosc de Montjuïc, Barcelona
  - Escola Ramon Casas, Barcelona
  - Escola Seat, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Only after finishing the study and with the express authorization of the Department of Education of the Generalitat of Catalonia, the data processed and anonymized will be stored in a specialized repository for research purposes. The data in this repository will be placed under the Creative Commons Attribution-Non Comercial-Share Alike (CC BY-NC-SA) license. They will only be used for scientific purposes and after requesting permission from the authors and under the same conditions that we have established. The following data will not be made publicly available:
  * Personal data and other data that can be tracked to participants identity.
  * Data that compromises the protection of a partner(s) intellectual property.
  * The level of data made available will also be considered, for example, pre-processed data will not be provided unless there is a clear reason for doing so.
  * Datasets which cannot be shared because of legal and contractual reasons.
Supporting Information: Study Protocol, SAP
Time Frame: After finishing the study
Access Criteria: Once processing, quality control, organisation, analysis, and publication are complete, the data will be made accessible by deposition in open access repositories (https://b2share.eudat.eu).
  Members of the research team will form a data access committee. This committee will oversee that openly accessible data respect ethical and data security aspects, including intellectual property requirements. The possibilities of accessing the data in the specialized repository will always be decided in consultation with our collaborators and the Department of Education of the Generalitat de Catalunya.

REFERENCES:
- [Background] Smits-Engelsman B, Verbecque E. Pediatric care for children with developmental coordination disorder, can we do better? Biomed J. 2022 Apr;45(2):250-264. doi: 10.1016/j.bj.2021.08.008. Epub 2021 Sep 2. PMID 34482014
- [Background] Adams IL, Lust JM, Wilson PH, Steenbergen B. Compromised motor control in children with DCD: a deficit in the internal model?-A systematic review. Neurosci Biobehav Rev. 2014 Nov;47:225-44. doi: 10.1016/j.neubiorev.2014.08.011. Epub 2014 Sep 1. PMID 25193246
- [Background] Fuster JM. Executive frontal functions. Exp Brain Res. 2000 Jul;133(1):66-70. doi: 10.1007/s002210000401. PMID 10933211
- [Background] Fuster JM. The prefrontal cortex in the neurology clinic. Handb Clin Neurol. 2019;163:3-15. doi: 10.1016/B978-0-12-804281-6.00001-X. PMID 31590737
- [Background] Goto K, Hoshi Y, Sata M, Kawahara M, Takahashi M, Murohashi H. Role of the prefrontal cortex in the cognitive control of reaching movements: near-infrared spectroscopy study. J Biomed Opt. 2011 Dec;16(12):127003. doi: 10.1117/1.3658757. PMID 22191933
- [Background] Jueptner M, Stephan KM, Frith CD, Brooks DJ, Frackowiak RS, Passingham RE. Anatomy of motor learning. I. Frontal cortex and attention to action. J Neurophysiol. 1997 Mar;77(3):1313-24. doi: 10.1152/jn.1997.77.3.1313. PMID 9084599
- [Background] Kumar N, Sidarta A, Smith C, Ostry DJ. Ventrolateral Prefrontal Cortex Contributes to Human Motor Learning. eNeuro. 2022 Sep 29;9(5):ENEURO.0269-22.2022. doi: 10.1523/ENEURO.0269-22.2022. Print 2022 Sep-Oct. PMID 36114001
- [Background] Hampshire A, Duncan J, Owen AM. Selective tuning of the blood oxygenation level-dependent response during simple target detection dissociates human frontoparietal subregions. J Neurosci. 2007 Jun 6;27(23):6219-23. doi: 10.1523/JNEUROSCI.0851-07.2007. PMID 17553994
- [Background] Passingham RE, Toni I, Rushworth MF. Specialisation within the prefrontal cortex: the ventral prefrontal cortex and associative learning. Exp Brain Res. 2000 Jul;133(1):103-13. doi: 10.1007/s002210000405. PMID 10933215
- [Background] Bunge SA, Kahn I, Wallis JD, Miller EK, Wagner AD. Neural circuits subserving the retrieval and maintenance of abstract rules. J Neurophysiol. 2003 Nov;90(5):3419-28. doi: 10.1152/jn.00910.2002. Epub 2003 Jul 16. PMID 12867532
- [Background] Blank R, Smits-Engelsman B, Polatajko H, Wilson P; European Academy for Childhood Disability. European Academy for Childhood Disability (EACD): recommendations on the definition, diagnosis and intervention of developmental coordination disorder (long version). Dev Med Child Neurol. 2012 Jan;54(1):54-93. doi: 10.1111/j.1469-8749.2011.04171.x. No abstract available. PMID 22171930
- [Background] Ferrer-Uris B, Busquets A, Angulo-Barroso R. Adaptation and Retention of a Perceptual-Motor Task in Children: Effects of a Single Bout of Intense Endurance Exercise. J Sport Exerc Psychol. 2018 Feb 1;40(1):1-9. doi: 10.1123/jsep.2017-0044. Epub 2018 Mar 9. PMID 29523049
- [Background] Angulo-Barroso R, Ferrer-Uris B, Busquets A. Enhancing Children's Motor Memory Retention Through Acute Intense Exercise: Effects of Different Exercise Durations. Front Psychol. 2019 Aug 28;10:2000. doi: 10.3389/fpsyg.2019.02000. eCollection 2019. PMID 31555181
- [Background] Kagerer FA, Bo J, Contreras-Vidal JL, Clark JE. Visuomotor adaptation in children with developmental coordination disorder. Motor Control. 2004 Oct;8(4):450-60. doi: 10.1123/mcj.8.4.450. PMID 15585900
- [Background] Kagerer FA, Contreras-Vidal JL, Bo J, Clark JE. Abrupt, but not gradual visuomotor distortion facilitates adaptation in children with developmental coordination disorder. Hum Mov Sci. 2006 Oct;25(4-5):622-33. doi: 10.1016/j.humov.2006.06.003. Epub 2006 Oct 2. PMID 17011655
- [Background] King BR, Kagerer FA, Harring JR, Contreras-Vidal JL, Clark JE. Multisensory adaptation of spatial-to-motor transformations in children with developmental coordination disorder. Exp Brain Res. 2011 Jul;212(2):257-65. doi: 10.1007/s00221-011-2722-z. Epub 2011 May 17. PMID 21584627
- [Background] Lundbye-Jensen J, Skriver K, Nielsen JB, Roig M. Acute Exercise Improves Motor Memory Consolidation in Preadolescent Children. Front Hum Neurosci. 2017 Apr 20;11:182. doi: 10.3389/fnhum.2017.00182. eCollection 2017. PMID 28473761
- [Background] Preston N, Magallon S, Hill LJ, Andrews E, Ahern SM, Mon-Williams M. A systematic review of high quality randomized controlled trials investigating motor skill programmes for children with developmental coordination disorder. Clin Rehabil. 2017 Jul;31(7):857-870. doi: 10.1177/0269215516661014. Epub 2016 Aug 1. PMID 27481937
- [Background] Smits-Engelsman BC, Wilson PH, Westenberg Y, Duysens J. Fine motor deficiencies in children with developmental coordination disorder and learning disabilities: an underlying open-loop control deficit. Hum Mov Sci. 2003 Nov;22(4-5):495-513. doi: 10.1016/j.humov.2003.09.006. PMID 14624830
- [Background] Wilmut K, Wann J. The use of predictive information is impaired in the actions of children and young adults with Developmental Coordination Disorder. Exp Brain Res. 2008 Dec;191(4):403-18. doi: 10.1007/s00221-008-1532-4. Epub 2008 Aug 16. PMID 18709366
- [Background] Wilson PH, Maruff P, Lum J. Procedural learning in children with developmental coordination disorder. Hum Mov Sci. 2003 Nov;22(4-5):515-26. doi: 10.1016/j.humov.2003.09.007. PMID 14624831
- [Background] Wilson PH, Ruddock S, Smits-Engelsman B, Polatajko H, Blank R. Understanding performance deficits in developmental coordination disorder: a meta-analysis of recent research. Dev Med Child Neurol. 2013 Mar;55(3):217-28. doi: 10.1111/j.1469-8749.2012.04436.x. Epub 2012 Oct 29. PMID 23106668
- [Background] Zwicker JG, Missiuna C, Harris SR, Boyd LA. Developmental coordination disorder: a review and update. Eur J Paediatr Neurol. 2012 Nov;16(6):573-81. doi: 10.1016/j.ejpn.2012.05.005. Epub 2012 Jun 15. PMID 22705270